CLINICAL TRIAL: NCT02441101
Title: Right Ventricular Septal Pacing in Patients With Right Bundle Branch Block and Heart Failure, a Pilot Clinical Trial (The SPARK Trial)
Brief Title: Right Ventricular Septal Pacing in Patients With Right Bundle Branch Block and Heart Failure (The SPARK Trial)
Acronym: SPARK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Barry London (Other)
Responsible Party: Sponsor-Investigator, Barry London, PI, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201409760
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Right Bundle-Branch Block; Heart Failure
Keywords: Cardiac Resynchronization therapy
MeSH Terms: conditions — Bundle-Branch Block; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RV pacing optimization on/off (Experimental): RBBB pacing Arm 1 is RV pacing optimization on/off
  Interventions: Device: RV DDD(R)-60 with AV optimization
- RV pacing optimization off/on (Placebo Comparator): Standard demand pacing Arm 2 is RV pacing optimization off/on
  Interventions: Device: RV DDD(R)-60

INTERVENTIONS:
Device: RV DDD(R)-60 with AV optimization — Device to be programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG
  Arms: RV pacing optimization on/off
Device: RV DDD(R)-60 — AV settings programmed to minimize RV pacing - standard demand pacing programming.
  Arms: RV pacing optimization off/on

SUMMARY:
This clinical study has been designed to test whether a new pacing therapy would lead to improvement in heart function, symptoms and quality of life in a specific group of heart failure patients. This group has a unique electrical conduction problem (Right Bundle Branch Block) that did not respond well to the current available pacing therapy.

DETAILED DESCRIPTION:
This pilot clinical trial will be a randomized single blinded cross over trial. Each subject will undergo three study stages. Subject will be randomized initially to either of the two arms; experimental or placebo, and then will be followed up for 3 months for the first stage to assess outcomes. In the second stage, both arms transition to a two months, intervention free, wash out period. Finally, at the third stage both arms will cross over and subject will be followed up for an additional 3 months for outcomes assessment.

ELIGIBILITY:
Inclusion Criteria:

* Cardiomyopathy; ischemic or non-ischemic on optimal medical therapy per current heart failure treatment guidelines for at least 3 months.
* LVEF < 35% by trans-thoracic echocardiogram assessment
* Prior implantation of pacemaker/defibrillator with at least an atrial and RV mid septal lead. Atrial lead can be waived if RV lead has atrial sensing capabilities*
* Normal sinus rhythm at enrollment
* RBBB with QRS duration >120 msec on 12 lead surface EKG.
* PR interval <250 msec on 12 lead surface EKG

  * Subjects with biventricular pacemaker/ICD will be eligible for enrollment if their LV lead pacing function has been turned off by the subject's primary cardiologist prior to study enrollment for at least 3 months (this could be due to lead malfunction or the decision to deactivate the LV pacing therapy for any reason per primary cardiologist discretion)

Exclusion Criteria:

* Age younger than 18 years old
* Pregnancy
* Acute Myocardial infarction within 6 months of entry into the study
* Inotrope dependent heart failure condition
* Left ventricular assist device or heart transplantation
* Any other known conditions other than heart failure that could limit survival to < 6 months.
* Atrial fibrillation or flutter burden >10% of the time within the last 6 months
* Atrioventricular node disease that requires ventricular pacemaker support >10% of the time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Giudici, MD, Study Chair — University of Iowa; Michael C Giudici, MD, Principal Investigator — University of Iowa; Shubba D Roy, MD, Principal Investigator — University of Iowa; Trisha Elliott, RTR, Study Director — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RV Pacing Optimization on First, Then Off: Arm 1 is RV pacing optimization on first, then off
  After baseline measurements, RV DDD(R)-60 with AV optimization (Device is programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG) is turned on for 3 months. After the outcome measurements, RV DDD(R)-60 with AV optimization is turned off for 3 months and final outcome measurements are performed. This is a crossover study.
- RV Pacing Optimization Off First, Then on: Arm 2 is RV pacing optimization off first then on
  After baseline measurements, RV DDD(R)-60 with AV optimization (Device is programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG) is turned off for 3 months. After the outcome measurements, RV DDD(R)-60 with AV optimization is turned on for 3 months and final outcome measurements are performed. This is a crossover study.
Period: Overall Study
Arm/Group | RV Pacing Optimization on First, Then Off | RV Pacing Optimization Off First, Then on
Started | 4 | 2
Completed | 1 | 2
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — PI relocated and study terminated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- RV Pacing Optimization on First, Then Off: RV Pacing Optimization on first, then Off
  RV DDD(R)-60 with AV optimization: Device to be programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG
- RV Pacing Optimization Off First, Then on: RV Pacing Optimization off first, then on
  RV DDD(R)-60: AV settings programmed to minimize RV pacing - standard demand pacing programming.
- Total: Total of all reporting groups
Arm/Group | RV Pacing Optimization on First, Then Off | RV Pacing Optimization Off First, Then on | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (9) | 62 (15) | 70 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change of LV Ejection Fraction Compared to Baseline
Description: LV Ejection Fraction is defined as [(end diastolic volume minus end systolic volume) / (end diastolic volume] as measured by echocardiography.
  Comparison of LV Ejection Fraction with RV pacing optimization on vs. RV pacing optimization off.
  Arm 1 is RV pacing optimization on then off Arm 2 is RV pacing optimization off then on
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- RV Pacing Optimization on: Arm 1 is RV pacing optimization on
  RV DDD(R)-60 with AV optimization: Device to be programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG
- RV Pacing Optimization Off: Arm 2 is RV pacing optimization off
  RV DDD(R)-60: AV settings programmed to minimize RV pacing - standard demand pacing programming.
Arm/Group | RV Pacing Optimization on | RV Pacing Optimization Off
Number analyzed (Participants) | 6 | 3
Percent | 0 (4) | 4 (7)

2. Secondary Outcome: Electrocardiographic: QRS Duration
Description: Comparing baseline to intervention on Comparing intervention off to intervention off Expect statistically significant decrease with intervention on
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- RV Pacing Optimization on: RV Pacing Optimization on
  RV DDD(R)-60 with AV optimization: Device to be programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG
- RV Pacing Optimization Off: RV Pacing Optimization off
  RV DDD(R)-60: AV settings programmed to minimize RV pacing - standard demand pacing programming.
Arm/Group | RV Pacing Optimization on | RV Pacing Optimization Off
Number analyzed (Participants) | 6 | 3
Milliseconds | -36 (22) | 2 (9)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected during enrollment period, up to 6 months
Description: Medical record review and directly from participants
Groups:
- RV Pacing Optimization on: Arm 1 RV pacing optimization on
  RV DDD(R)-60 with AV optimization: Device to be programmed for RV pacing with AV interval optimization at the bedside to produce QRS fusion with the native conduction down the native left bundle on surface EKG
Arm/Group | RV Pacing Optimization on | RV Pacing Optimization Off
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-12-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02441101/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02441101/SAP_001.pdf